CLINICAL TRIAL: NCT04693260
Title: A Clinical Study to Evaluate the Remote Monitoring of Myopia Patients With the EyeQue Insight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EyeQue Corp. (Industry)
Collaborators: Eye Boutique Optometry (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: EYEQUE - 007
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Myopia
Keywords: myopia; Ortho-k; vision
MeSH Terms: conditions — Myopia | interventions — Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hand-held Device Supported by Mobile Application (Other): Insight device ETDRS measurement compared to a standard ETDRS chart
  Interventions: Device: Visual Acuity with a Hand-held Device Supported by Mobile App.

INTERVENTIONS:
Device: Visual Acuity with a Hand-held Device Supported by Mobile App. — The Insight will be compared to a standard ETDRS eyechart

SUMMARY:
The objective of this study is to determine whether the remote monitoring of myopia patients with the EyeQue Insight (visual acuity test) can replace regularly scheduled follow-up visits.

DETAILED DESCRIPTION:
A prospective exploratory study to determine whether the remote monitoring of myopia patients with the EyeQue Insight (visual acuity test) can replace regularly scheduled follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Ages =>7 y.o.
3. Subjects that are minors (<18 years old) must have a parent or legal guardian.
4. Binocular vision
5. Willing and able to give informed consent and follow all study procedures and requirements
6. Fluent in English
7. Be treated for myopia with Ortho-K, day contacts, or night contacts

Exclusion Criteria:

1. Has been diagnosed within 4 weeks, or currently has signs or symptoms, of COVID-19.
2. Has traveled outside the country within the last 4 weeks
3. Medications:

   a. Taking medications that may affect ability to follow instructions.
4. Eye Disease:

   a. Subjects with eye disease deemed by the Investigator to be inappropriate for the study such as an active eye infection, keratoconus, etc.
5. Subjects that:

   1. Lack physical dexterity to properly operate the EyeQue App on the smartphone
   2. Lack the ability to follow instruction
   3. Lack binocular vision
   4. Lack the ability to maintain both eyes open
   5. Had eye surgery within the last 12 months (including Lasik)

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Departure from scheduled follow-up visits with clinical confirmation | Approximately 21 Weeks
  Site will monitor the patient remotely and determine if the subject should depart from their scheduled visits based on at-home testing. If visit departure is warranted the site will examine them in the office and confirm if a departure from normally schedule visit was warranted.

SECONDARY OUTCOMES:
Measure rapidly changing visual acuity | Approximately 21 Weeks
  Ability to track and measure visual acuity with the EyeQue Insight in patients with rapidly changing visual acuity during the first month of Ortho-K introduction.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Boutique Optometry, Santa Clara, California, United States

IPD SHARING:
Plan to Share IPD: No